CLINICAL TRIAL: NCT01482520
Title: Genome-wide Association Study to Predict Treatment Response for Molecular Targeted Therapy in Hepatocellular Carcinoma and Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: 2008-06-050
Record Dates: First submitted 2011-11-14; First posted 2011-11-30 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Hepatocellular Carcinoma; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Renal cell carcinoma
- Hepatocellular carcinoma patients

SUMMARY:
All Hepatocellular carcinoma and Renal cell carcinoma patients who receive molecular targeted therapy will be candidates for the study.

No additional treatment or intervention will be conducted except for blood sampling that will be limited to one time only.

Blood samples (10 cc in volume) will be collected from all study participants once they provided written informed consent form. DNA will be extracted from peripheral blood samples using DNA isolation kit.

ELIGIBILITY:
Inclusion Criteria:

* All Hepatocellular carcinoma and Renal cell carcinoma patients who receive molecular targeted therapy will be candidates for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Hepatocellular carcinoma and Renal cell carcinoma patients who receive molecular targeted therapy will be candidates for the study.
  Once the patient signed written informed consent, two bottles of 5 cc blood will be drawn and subsequently extracted DNA and serum will be stored until genetic analysis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Genotypes | 36months
  To define genotypes of HCC and RCC patients who will likely to response to molecular targeted therapy.
  To define genotypes associated with adverse events from molecular targeted.
  To identify genotypes which will predict survival or disease-free survival following molecular targeted therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea